CLINICAL TRIAL: NCT04126733
Title: An Open-label, Single-arm, Phase II Study of Regorafenib and Nivolumab in Patients With Mismatch Repair-Proficient (pMMR)/Microsatellite Stable (MSS) Colorectal Cancer (CRC)
Brief Title: Study on the Effectiveness and Safety of the Combination of the Two Drugs Regorafenib and Nivolumab in Patients With Colorectal Cancer (Cancer of the Colon or Rectum Classified as Proficient Mismatch Repair and Microsatellite Stable)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20975
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib + Nivolumab (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Biological: Nivolumab (Opdivo)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Regorafenib administered as oral tablets given every day for 3 weeks of each 28 days treatment cycle (i.e., 3 weeks on, 1 week off)
Biological: Nivolumab (Opdivo) — Administered on day 1 of every treatment cycle.

SUMMARY:
The purpose of this study is to learn if combination of the two drugs regorafenib and nivolumab is an effective treatment for pMMR - MSS colorectal cancer, a special type of cancer of the colon or rectum (pMMR stands for proficient Mismatch Repair; MSS stands for Microsatellite Stable) and whether it is safe for patients. Regorafenib works by blocking several different proteins involved in tumor growth. Nivolumab is an immunotherapy drug encouraging the body's own immune system to attack cancer cells.

Both drugs have been approved, but not for how they are being used as combination therapy in this study. Brand name of regorafenib is Stivarga; brand name of nivolumab is Opdivo.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed advanced, metastatic, or progressive pMMR/MSS adenocarcinoma of colon or rectum
* Participant must have progressed or be intolerant to prior systemic chemotherapy including fluoropyrimidines, irinotecan, oxaliplatin, anti-vascular endothelial growth factor (VEGF) therapy, and, if extended rat sarcoma viral oncogene homolog (RAS) wild type, an anti-epidermal growth factor receptor (EGFR) therapy. Exceptions may apply
* Participants must have adequate organ and marrow function defined by protocol-specified laboratory tests
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Measurable disease as determined by response evaluation criteria in solid tumors (RECIST) v1.1
* Provision of recently obtained tumor tissue as per protocol specified requirement
* Anticipated life expectancy greater than 3 months
* Be able to swallow and absorb oral tablets

Exclusion Criteria:

* Participants with Mismatch repair deficient (dMMR) / microsatellite instable-high (MSI-H) colorectal cancer
* Prior therapy with regorafenib, anti-programmed cell death protein 1 (PD-1), programmed cell death protein 1 ligand 1 (PD-L1), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors, or any form of immunotherapy to treat cancer
* Presence of active central nervous system (CNS) metastases; participants with stable CNS disease or previously treated lesions are eligible for study entry
* Poorly controlled hypertension, defined as a blood pressure consistently above 150/90 mmHg despite optimal medical management
* Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within 6 months before the start of study medication. Active pulmonary emboli or deep vein thrombosis that are significant or not adequately controlled on anticoagulation regimen
* Any hemorrhage or bleeding event ≥ National Cancer Institute - Common terminology criteria for adverse events (NCI-CTCAE) Grade 3 within 28 days prior to the start of study medication
* Participants with an active, known or suspected autoimmune disease
* History of interstitial lung disease or pneumonitis
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection
* Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Miami Cancer Institute at Baptist Health South Florida, Miami, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Nebraska Cancer Specialists, Papillion, Nebraska
  - New York Oncology Hematology. P.C., Albany, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology-Arlington North, Arlington, Texas
  - Baylor Charles A. Sammons Cancer Center at Dallas, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - Virginia Oncology Associates, Newport News, Virginia
  - Northwest Cancer Specialists, PC, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Fakih M, Raghav KPS, Chang DZ, Larson T, Cohn AL, Huyck TK, Cosgrove D, Fiorillo JA, Tam R, D'Adamo D, Sharma N, Brennan BJ, Wang YA, Coppieters S, Zebger-Gong H, Weispfenning A, Seidel H, Ploeger BA, Mueller U, Oliveira CSV, Paulson AS. Regorafenib plus nivolumab in patients with mismatch repair-proficient/microsatellite stable metastatic colorectal cancer: a single-arm, open-label, multicentre phase 2 study. EClinicalMedicine. 2023 Apr 6;58:101917. doi: 10.1016/j.eclinm.2023.101917. eCollection 2023 Apr. PMID 37090438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 12 centers (of which at least one participant was treated) in the United States between 14-OCT-2019 (first participant first visit) and 28-MAR-2022 (last participant last visit).
Pre-assignment Details: A total of 94 participants were screened to enter the study; 21 participants were screening failures and 3 participants discontinued before completion of screening (2 participants withdrew consent and 1 participant died during screening). A total of 70 participants were assigned to treatment and received at least one dose of study treatment.
Groups:
- Regorafenib Plus Nivolumab: Regorafenib was administrated 2x40 mg once daily (q.d.) on cycle 1 and up to 3x40 mg q.d. from cycle 2 onward for 3 weeks of each 28 days treatment cycle (21 days on/7 days off).
  Nivolumab was administrated 480 mg on day 1 of each 28 days treatment cycle (Q4W).
Period: Treatment Period
Arm/Group | Regorafenib Plus Nivolumab
Started | 70
Completed | 0
Not Completed | 70
Not completed — Progressive Disease - Radiological Progression | 47
Not completed — Adverse Event | 8
Not completed — Progressive Disease - Clinical Assessment | 7
Not completed — Physician Decision | 5
Not completed — Death | 1
Not completed — Other Reasons | 2
Period: Active Follow-up Period
Arm/Group | Regorafenib Plus Nivolumab
Started | 39 (Participants had the option to decline participation in active follow-up.)
Completed | 19
Not Completed | 20
Not completed — Death | 13
Not completed — Progressive Disease - Clinical Assessment | 4
Not completed — Withdrawal by Subject | 2
Not completed — Other Reasons | 1
Period: Long-term Follow-up Period
Arm/Group | Regorafenib Plus Nivolumab
Started | 29 (All participants who accepted long-term follow-up.)
Completed | 0
Not Completed | 29
Not completed — Death | 22
Not completed — Withdrawal by Subject | 1
Not completed — Ongoing with Long Term Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 10
  White | 50
  More than one race | NA — This category was not investigated.
  Unknown or Not Reported | 2
Baseline ECOG Performance Status [Number; unit: participants] — The participant's ability to manage activities of daily living at baseline was appraised utilizing the performance status scale by Eastern Cooperative Oncology Group (ECOG).
  Grade 0: Fully active, able to carry on all pre-diseases performance without restriction.
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  participants
    0 - Fully Active | 36
    1 - Restricted Activity | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 Assessed by Investigator
Description: ORR was defined as the percentage of participants with overall response of complete response (CR) or partial response (PR).
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have decreased in size to have a short axis of < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: Through database cut-off date of 11-NOV-2020 (Primary Completion Date) (up to 13 months)
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage (%) of participants
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 70
percentage (%) of participants | 7.1 [2.4 to 15.9]
Statistical Analysis 1: Comparison: Regorafenib Plus Nivolumab; Test type: Equivalence — H0: ORR ≤ 5% versus H1: ORR >5% The hypothesis was tested by a one-sided exact binomial test, assuming a background response rate for the combination to be at most 5%; p = 0.2721, Exact Binomial Test — The target response rate for the combination treatment was 17%. Using a one-sided exact binomial test at a type-I error of at most 2.5% at least 8 responders out of the 70 patients were needed to achieve significance; Rate = 7.1, 95% CI [2.4 to 15.9]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined for responders only as the time from first documentation of response (i.e. CR or PR) until disease progression or death (if death without documented disease progression).
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have decreased in size to have a short axis of < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: Through last patient last visit (LPLV) at date of 28 MAR 2022 (up to 30 months)
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 5
weeks | NA [16.14 to NA] — Median, upper bound for 95% confidence interval could not be calculated due to insufficient number of participants with event.

3. Secondary Outcome: Disease Control Rate (DCR) at 8 and 16 Weeks
Description: DCR was defined as the percentage of participants with tumor response of complete response (CR), partial response (PR) or stable disease (SD).
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have decreased in size to have a short axis of < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: At 8, 16, 24, 32 and 40 weeks
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage (%) of participants
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 70
percentage (%) of participants
  Disease Control Rate at 8 weeks | 38.6 [27.2 to 51.0]
  Disease Control Rate at 16 weeks | 38.6 [27.2 to 51.0]
  Disease Control Rate at 24 weeks | 38.6 [27.2 to 51.0]
  Disease Control Rate at 32 weeks | 38.6 [27.2 to 51.0]
  Disease Control Rate at 40 weeks | 38.6 [27.2 to 51.0]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was the time from first dose of study medication to disease progression or death, whichever was earlier.
Time Frame: Through last patient last visit (LPLV) at date of 28 MAR 2022 (up to 30 months)
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 70
weeks | 8.00 [7.86 to 10.57]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from first dose of the study treatment to death. For patients who did not die, OS was censored at the last time point at which the survival status was known to be alive.
Time Frame: Through last patient last visit (LPLV) at date of 28 MAR 2022 (up to 30 months)
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 70
weeks | 51.86 [30.29 to 69.71]

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Different Severity Types of TEAEs Per Common Terminology Criteria for Adverse Events (CTCAE) v5
Description: TEAEs were started during treatment or within the post-treatment time window (30 days after last dose of regorafenib and 100 days after last dose of nivolumab.).
  TEAEs were summarized by system organ class (SOC) and preferred term, severity (based on CTCAE v5 grades). Laboratory data considered as AE were graded according to CTCAE v5.
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: 30 days after last dose of regorafenib and 100 days after last dose of nivolumab until study completion (up to 30 months)
Population: Full Analysis Set (FAS)
Measure: Number; unit: participants
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 70
participants
  Any AEs | 69
  Serious AEs | 34
  Worst grade: Grade 1 | 3
  Worst grade: Grade 2 | 18
  Worst grade: Grade 3 | 38
  Worst grade: Grade 4 | 7
  Worst grade: Grade 5 (death) | 3
  Worst grade: Grade 1 or 2 | 21
  Worst grade: Grade 3 or 4 | 45
  Worst grade: Grade 3, 4, or 5 | 48
  Grade 5 (death) between Day X+1 and Day 30 | 3
  Grade 5 (death) between Day 31 and Day 100 | 0

7. Post Hoc Outcome: Duration of Stable Disease
Description: Duration of stable disease was measured from the start of the treatment until the criteria for progression were met.
Time Frame: Through last patient last visit (LPLV) at date of 28 MAR 2022 (up to 30 months)
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Regorafenib Plus Nivolumab
Number analyzed (Participants) | 22
weeks | 29.86 [15.86 to 32.00]

ADVERSE EVENTS:
Time Frame: An adverse event (AE) was considered as treatment-emergent (TEAE) if it started during treatment or within the post-treatment time window (30 days after last dose of regorafenib and 100 days after last dose of nivolumab) until study completion (up to 30 months).
Groups:
- Regorafenib Plus Nivolumab: Regorafenib was administrated 2x40mg q.d. (cycle 1) then up to 3x40mg q.d. (from cycle 2 onward) for 3 weeks of each 28 days treatment cycle. Nivolumab was administrated 480mg on day 1 of each 28 days treatment cycle.
Arm/Group | Regorafenib Plus Nivolumab
All-Cause Mortality (participants affected / at risk) | 40/70
Serious Adverse Events (participants affected / at risk) | 34/70
Other Adverse Events (participants affected / at risk) | 66/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Plus Nivolumab (N=70)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (4)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pyelonephritis (Infections and infestations) | 1 (3)
Sepsis (Infections and infestations) | 4 (5)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urosepsis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (4)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pyelonephritis (Infections and infestations) | 1 (3)
Sepsis (Infections and infestations) | 4 (5)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urosepsis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (4)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Pyelonephritis (Infections and infestations) | 1 (3)
Sepsis (Infections and infestations) | 4 (5)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urosepsis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Plus Nivolumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 13 (24)
Hypothyroidism (Endocrine disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 15 (18)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9)
Constipation (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 14 (18)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 16 (18)
Stomatitis (Gastrointestinal disorders) | 11 (13)
Vomiting (Gastrointestinal disorders) | 12 (16)
Asthenia (General disorders) | 4 (4)
Chills (General disorders) | 6 (7)
Fatigue (General disorders) | 30 (50)
Malaise (General disorders) | 4 (8)
Mucosal inflammation (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 6 (7)
Pyrexia (General disorders) | 16 (22)
Bronchitis (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 10 (12)
Alanine aminotransferase increased (Investigations) | 12 (17)
Aspartate aminotransferase increased (Investigations) | 13 (18)
Blood bilirubin increased (Investigations) | 17 (32)
Blood lactate dehydrogenase increased (Investigations) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (9)
Lipase increased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 6 (13)
Weight decreased (Investigations) | 11 (18)
Blood alkaline phosphatase increased (Investigations) | 10 (15)
Dehydration (Metabolism and nutrition disorders) | 9 (14)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (11)
Decreased appetite (Metabolism and nutrition disorders) | 21 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Dizziness (Nervous system disorders) | 4 (7)
Headache (Nervous system disorders) | 11 (15)
Proteinuria (Renal and urinary disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (29)
Hypertension (Vascular disorders) | 11 (14)
Hypotension (Vascular disorders) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 13 (24)
Hypothyroidism (Endocrine disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 15 (18)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9)
Constipation (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 14 (18)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 16 (18)
Stomatitis (Gastrointestinal disorders) | 11 (13)
Vomiting (Gastrointestinal disorders) | 12 (16)
Asthenia (General disorders) | 4 (4)
Chills (General disorders) | 6 (7)
Fatigue (General disorders) | 30 (50)
Malaise (General disorders) | 4 (8)
Mucosal inflammation (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 6 (7)
Pyrexia (General disorders) | 16 (22)
Bronchitis (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 10 (12)
Alanine aminotransferase increased (Investigations) | 12 (17)
Aspartate aminotransferase increased (Investigations) | 13 (18)
Blood bilirubin increased (Investigations) | 17 (32)
Blood lactate dehydrogenase increased (Investigations) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (9)
Lipase increased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 6 (13)
Weight decreased (Investigations) | 11 (18)
Blood alkaline phosphatase increased (Investigations) | 10 (15)
Dehydration (Metabolism and nutrition disorders) | 9 (14)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (11)
Decreased appetite (Metabolism and nutrition disorders) | 21 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Dizziness (Nervous system disorders) | 4 (7)
Headache (Nervous system disorders) | 11 (15)
Proteinuria (Renal and urinary disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (29)
Hypertension (Vascular disorders) | 11 (14)
Hypotension (Vascular disorders) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 13 (24)
Hypothyroidism (Endocrine disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 15 (18)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9)
Constipation (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 14 (28)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 17 (21)
Stomatitis (Gastrointestinal disorders) | 11 (13)
Vomiting (Gastrointestinal disorders) | 12 (17)
Asthenia (General disorders) | 4 (4)
Chills (General disorders) | 6 (7)
Fatigue (General disorders) | 30 (50)
Malaise (General disorders) | 4 (8)
Mucosal inflammation (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 4 (5)
Pyrexia (General disorders) | 16 (22)
Bronchitis (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 11 (13)
Alanine aminotransferase increased (Investigations) | 12 (17)
Aspartate aminotransferase increased (Investigations) | 13 (18)
Blood bilirubin increased (Investigations) | 17 (32)
Blood lactate dehydrogenase increased (Investigations) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (9)
Lipase increased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 6 (13)
Weight decreased (Investigations) | 11 (18)
Blood alkaline phosphatase increased (Investigations) | 10 (15)
Dehydration (Metabolism and nutrition disorders) | 9 (14)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (11)
Decreased appetite (Metabolism and nutrition disorders) | 21 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Dizziness (Nervous system disorders) | 4 (7)
Headache (Nervous system disorders) | 11 (15)
Proteinuria (Renal and urinary disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (29)
Hypertension (Vascular disorders) | 11 (14)
Hypotension (Vascular disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Preliminary efficacy assessment suggested that the study would not meet its primary efficacy endpoint, therefore the study was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may publish or present individual study data (including case reports) obtained in the course of this study but only after the primary report and/or publication of the study results in their entirety. If publishing individual site data is foreseen, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04126733/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT04126733/SAP_001.pdf